CLINICAL TRIAL: NCT06471075
Title: Brief (i.e., <10 Minute) Behavioral Intervention for Pain
Brief Title: Brief Mindfulness Intervention for Pain Before an In-clinic Orthopedic Procedure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00004916
Record Dates: First submitted 2024-06-13; First posted 2024-06-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Pain; Chronic Pain; Acute Pain
Keywords: mindfulness; kyphoplasty; radiofrequency ablation
MeSH Terms: conditions — Pain; Chronic Pain; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Pain Management (Experimental)
  Interventions: Behavioral: Mindful Pain Management
- Pain Psychoeducation (Active Comparator)
  Interventions: Behavioral: Pain Psychoeducation

INTERVENTIONS:
Behavioral: Mindful Pain Management — The mindfulness intervention will involve a 2-minute introduction to mindfulness as a technique for pain management followed by a 5-minute, audio-guided, mindful breathing practice.
  Arms: Mindfulness Pain Management
Behavioral: Pain Psychoeducation — In the pain psychoeducation intervention, participants will be provided timematched information about different pain management strategies (e.g., ice, rest) and accessible resources to promote overall well-being.
  Arms: Pain Psychoeducation

SUMMARY:
This project is a single-site, randomized controlled trial designed to investigate the impact of a 7-minute mindfulness intervention on pain among patients undergoing kyphoplasty or radiofrequency ablation.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Kyphoplasty or Radiofrequency Ablation at Tallahassee Orthopedic Center
* Fluency with English
* Being 18 and above

Exclusion Criteria:

* Unable to consent because of physical or mental incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-22 (Actual); Primary Completion 2026-09-11 (Estimated); Study Completion 2026-09-11 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Unpleasantness Numeric Rating Scale | Immediately before to after 7-minute audio recording
  Change in acute pain unpleasantness will be measured with an individual item ("How unpleasant is your pain, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain unpleasantness.

SECONDARY OUTCOMES:
Acute Pain | Immediately before to after 7-minute audio recording
  Change in acute pain intensity will be measured with an individual item ("How much pain do you have, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain intensity.
Anxiety | Immediately before to after 7-minute audio recording
  Change in anxiety from baseline will be assessed with the Generalized Anxiety Disorder 2-item. Scores range from 0 to 6, with higher scores reflecting greater anxiety.
Treatment Satisfaction | At the end of the medical provider visit - approximately 1 hour.
  Treatment satisfaction at the visit's end will be measured with three, validated items (1. How satisfied are you with your medical care today?, 2. Was the visit/procedure tolerable?, 3. Would you have the same procedure again?), each scored on an 11-point, Likert-type scale ranging from 0 to 10. Higher scores represent greater treatment satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Tallahassee Orthopedic Clinic (TOC), Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No